CLINICAL TRIAL: NCT01465646
Title: Bioavailability Investigations of Thyronajod Mite Tablets of Dosage Strengths 50 μg Levothyrox-ine/75 μg Iodine, and 100 μg Levothyroxine/75 μg Iodine vs. a Levothyroxine Drinking-Solution: A Randomised Cross Over Study in Healthy Male Individuals. Currently: 100 μg/ 75 μg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Principal Investigator, Gerd Mikus, Head of Clinical Research Unit, Heidelberg University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: K069-2
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Pharmacokinetics
Keywords: levothyroxine; bioavailability
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- with idodine (Active Comparator)
  Interventions: Drug: levothyroxine
- without iodine (Experimental)
  Interventions: Drug: levothyroxine

INTERVENTIONS:
Drug: levothyroxine
  Arms: with idodine
Drug: levothyroxine
  Arms: without iodine

SUMMARY:
The purpose of this study is to measure the area under the curve (AUC0-48h; extent of systemic availability) and the maxi-mum concentrations (Cmax) of total serum levothyroxine (TT4, bound and free fraction) after a single pharmacological dose of 600 μg administered as tablets also containing iodine supple-ments vs. the same dose of levothyroxine administered as a reference solution without iodine.

ELIGIBILITY:
Inclusion Criteria:

* Euthyroid men
* Age: 18 - 50
* Normal values for fT4 und TSH
* Good state of health

Exclusion Criteria:

* Thyroid function disorders in terms of subclinical or overt hyper- or hypothyroidism
* History of thyroid function disorders
* Focal or diffuse autonomies of the thyroid gland
* Thyroid nodules >1 ml according to sonographic examination
* Any acute or chronic illness
* Dermatitis herpetiformis

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2003-06; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Unit, University of Heidelberg, Heidelberg, Germany